CLINICAL TRIAL: NCT05705531
Title: Assessment of Clonal Hematopoiesis and Its Relationship to Cardiovascular Disease in Hodgkin Lymphoma Survivors
Brief Title: A Study About How Blood Cell Growth Patterns Relate to Heart Health After Treatment for Hodgkin Lymphoma
Status: Recruiting | Type: Observational
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Other Study IDs: ALTE21C1; NCI-2022-09972 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ALTE21C1 (Other: Children's Oncology Group); COG-ALTE21C1 (Other: DCP); ALTE21C1 (Other: CTEP); UG1CA189955 (NIH)
Record Dates: First submitted 2023-01-11; First posted 2023-01-30 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Cardiovascular Disorder; Classic Hodgkin Lymphoma; Clonal Hematopoiesis
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational (blood samples, surveys, MRI, record review): Patients undergo collection of blood samples, complete surveys, and undergo cardiac MRI on study. Patients also have their medical records reviewed and may have archived blood samples collected if available.
  Interventions: Procedure: Archive Sample Retrieval; Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Procedure: Magnetic Resonance Imaging; Other: Survey Administration

INTERVENTIONS:
Procedure: Archive Sample Retrieval — Undergo collection of archived blood sample
  Other Names: ARCHIVE RETRIEVING
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Electronic Health Record Review — Undergo medical record abstraction
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Survey Administration — Complete surveys

SUMMARY:
This study assesses how blood cell growth patterns (clonal hematopoiesis) relate to heart health or cardiovascular disease (CVD) after treatment in patients with Hodgkin lymphoma. In some patients, cancer treatment at a young age may lead to later complications, including problems with heart health. Checking for blood cell growth patterns called therapy-related clonal hematopoiesis (t-CH) can help predict who might be at risk for heart health problems after Hodgkin lymphoma treatment. If doctors know who may be at greater risk for developing later heart complications, then they can more closely monitor those patients to prevent or detect heart complications early.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the prevalence of therapy-related clonal hematopoiesis (t-CH) possessing somatic mutations associated with cardiovascular disease (CVD) in anthracycline exposed pediatric classical Hodgkin Lymphoma patients detected after front line Hodgkin Lymphoma therapy.

II. To compare rates of t-CH possessing somatic mutations associated with CVD between anthracycline exposed pediatric classical Hodgkin Lymphoma patients with versus without objective signs of CVD according to cardiac magnetic resonance imaging (MRI).

SECONDARY OBJECTIVES:

I. To evaluate whether the incidence of t-CH possessing somatic mutations associated with CVD increases over time among pediatric classical Hodgkin Lymphoma patients previously treated with anthracyclines.

II. To compare rates of objective findings of CVD between groups of anthracycline exposed pediatric classical Hodgkin Lymphoma patients with versus without clinical risk factors for CVD.

EXPLORATORY OBJECTIVES:

I. To compare the prevalence of t-CH with mutations associated with CVD between anthracycline exposed pediatric classical Hodgkin Lymphoma patients who received versus did not receive mediastinal radiation as part of their initial treatment.

II. To assess whether specific patient characteristics and other treatment components (age, sex, race, dexrazoxane usage, etc.) are associated with an increased likelihood of t-CH with mutations associated with CVD.

III. To evaluate the effect of t-CH with mutations associated with CVD on objective findings of CVD, as adjusted for or mediated by other factors such as patient characteristics and clinical conditions associated with an elevated risk for CVD.

OUTLINE: This is an observational study.

Patients undergo collection of blood samples, complete surveys, and undergo cardiac MRI on study. Patients also have their medical records reviewed and may have archived blood samples collected if available.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be >= 7 years of age at the time of enrollment (age to perform an MRI without sedation).
* History of pathologically confirmed classical Hodgkin Lymphoma (cHL) initially diagnosed when the patient was >= 2 and < 22 years of age.
* As part of frontline therapy for cHL, the patient must have received a cumulative doxorubicin equivalent anthracycline dose of ≥ 200 mg/m^2 as estimated in doxorubicin isotoxic equivalents dose conversion calculation.

  * Note: History of COG therapeutic trial participation is not required. Institutional records (e.g., clinic note, treatment summary, chemotherapy roadmap) can be used as reference documentation of receipt of anthracycline dose.
* All systemic cancer treatment must have been completed ≥ 2 years prior to study enrollment.
* Not known to have had a primary event (relapse/second malignancy/death).

  * Note: Subjects treated at another institution are eligible if they are now being followed at the current COG institution, if the study procedures can be performed and the data accessible by a COG institution where the study is open.
* Patient must have access to cardiac MRI at the enrolling institution and must be able to complete cardiac MRI without sedation.

Exclusion Criteria:

* Medical contraindication to undergoing a non-contrast cardiac MRI.
* Patients with nodular lymphocyte-predominant HL.
* Received cancer therapy in addition to that for primary Hodgkin Disease (e.g., for disease progression or recurrence, or subsequent malignant neoplasm).
* History of CTCAE grade 3 or higher cardiovascular disease or condition known to exist prior to the patient's initial diagnosis of cHL.

  * Note: exceptions are made for congenital conditions considered fully resolved by surgery and chronic conditions such as hypertension or hypercholesterolemia that are managed with medical intervention.
* History of an immunodeficiency that existed prior to cHL diagnosis, such as primary immunodeficiency syndromes, organ transplant recipients and conditions requiring systemic immunosuppressive agents.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pathologically confirmed classical Hodgkin Lymphoma (cHL) initially diagnosed when the patient was >= 2 and < 22 years of age
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Therapy-related clonal hematopoiesis (t-CH) with mutations associated with cardiovascular disease | Up to 1 year
  Measured in the blood of eligible participants who were previously treated with anthracycline-containing therapy for pediatric classical Hodgkin lymphoma.

SECONDARY OUTCOMES:
Expansion of CH | Up to 1 year
  The outcome is the expansion of the CH, which will be expressed as the variant allele fraction (VAF) (CH verses the total normal DNA in the sample). Graphic analysis to reveal the time varying trend in the association between the expansion of CH over time and the presence/worsening of CVD signs and apply generalized estimating equation method (with each patient as cluster unit) to quantify this association while controlling for the potential correlation of repeated measurements within each patient.
Association between the presence of CVD and individual variables | Up to 1 year
  The outcome is the presence of CVD. This aim is to determine if there is an association between the presence of CVD and the individual variables constituting the clinical profile, either parametric (e.g., independent t-test, Chi^2-test, Pearson correlation coefficients) or nonparametric (e.g., Wilcoxon rank sum tests, Spearman's rank correlation coefficients) methods will be applied. Bootstrapping techniques might be used as a method of inference which does not rely on a specific underlying distribution. The statistical significance level will be set to 0.05 and all data analysis will be done using SAS statistical software (version 9.4).

OTHER OUTCOMES:
Prevalence and nature of CVD, CH and CH with mutations associated with cardiovascular disease | Up to 1 year
  The outcome is the expansion of the CH, which will be expressed as the variant allele fraction (VAF) (CH verses the total normal DNA in the sample). The VAFs and their exact 90% (Clopper-Pearson) confidence intervals are used to summarize the prevalence and nature of CVD, CH and CH with mutations associated with CVD for patients receiving mediastinal radiation.
Patient characteristics and treatments | Up to 1 year
  The outcome here is the incidence of t-CH with mutation. The specific patient characteristic and treatments (age, sex, race, dexrazoxane usage etc.) will be used to predict the incidence of t-CH with mutation rate. Regression model will be constructed to evaluate the effect of these patient characteristics and treatments on the incidence of t-CH with mutation rate, which will be presented by p-values, coefficients and their confidence intervals.
Effect of therapy-related clonal hematopoiesis on cardiovascular disease | Up to 1 year
  The outcome is the cardiovascular disease defined by cMRI. This aim is to evaluate the effect of other covariates such as patient characteristics (age, sex, race, etc.) and clinical conditions (radiation treatment with cardiac dosimetry, follow-up duration, etc.) on cardiovascular disease.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Hayashi, Principal Investigator — Children's Oncology Group
Locations (29):
- United States (28):
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Castellino SM, Giulino-Roth L, Harker-Murray P, Kahn JM, Forlenza C, Cho S, Hoppe B, Parsons SK, Kelly KM; COG Hodgkin Lymphoma Committee. Children's Oncology Group's 2023 blueprint for research: Hodgkin lymphoma. Pediatr Blood Cancer. 2023 Sep;70 Suppl 6(Suppl 6):e30580. doi: 10.1002/pbc.30580. Epub 2023 Jul 28. PMID 37505794